CLINICAL TRIAL: NCT04464252
Title: Development and Validation of an Automated Three-dimensional Cephalometry Method
Acronym: AutoCEPH-3D
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Laboratoire de Biomécanique Georges Charpak (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200215
Record Dates: First submitted 2020-06-17; First posted 2020-07-09 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Orthognathic Surgery; Dentofacial Deformities
Keywords: Imaging, three-dimensional; Cephalometry; Anatomic Landmarks; Radiographic Image Interpretation; Deep Learning; Orthodontics
MeSH Terms: conditions — Dentofacial Deformities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is aimed to develop and assess the validity of an algorithm for automated three-dimensional cephalometry.

DETAILED DESCRIPTION:
Cephalometric analysis is a standardized diagnostic method used daily by orthodontists and maxillofacial surgeons. It is based on linear and angular measurements performed on radiographic images. This examination is traditionally done manually on two-dimensional radiographs, which does not allow to analyze finely the bilateral structures which are found superimposed. Cephalometric analysis of three-dimensional imaging (cone beam computed tomography (CBCT) or computed tomography scan (CT-Scan)) may provide additional diagnostic information, particularly for patients with maxillofacial abnormalities or marked asymmetries.

One of the obstacle to the clinical use of three-dimensional cephalometric analysis is the time and expertise needed to manually place the landmarks. Automatic methods described in literature are preliminary and lack validation in a clinical context.

Our retrospective observational study is aimed to develop and validate a new automated three-dimensional cephalometry method. This method will be based on a deep learning algorithm trained from a database of pre-surgery CT-Scans of patients with have undergone an orthognathic surgery. These CT-Scans will be manually annotated to provide a reference standard for the training of the algorithm and its evaluation. The validation of our results will focus on demonstrating the diagnostic effectiveness and robustness of three-dimensional cephalometric measurements obtained in this clinical context.

ELIGIBILITY:
Inclusion Criteria:

1. Patients followed in the maxillofacial surgery department of Pitie-Salpetriere hospital (AP-HP, Paris, France) since 2014;
2. who underwent orthognathic surgery;
3. who had, for surgery planning, a three-dimensional radiographic examination (CT-Scan) which has been segmented for the manufacture of a custom-made device;
4. who did not object to the research.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care hospital (hopital de la Pitié-Salpêtrière, AP-HP, Paris, France), maxillofacial surgery department
Sampling Method: Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Average distances (in mm) between the points placed automatically and the points placed manually (reference). | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Percentage of points placed automatically within 2 / 3 / 4 mm of the the points placed manually (reference) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Maxillo-Faciale, Service de Chirurgie Maxillo-Faciale, Paris, France

IPD SHARING:
Plan to Share IPD: No